CLINICAL TRIAL: NCT03777696
Title: A Randomized Controlled Trial Comparing Co-administered Buccal Misoprostol and Intravenous Tranexamic Acid, Versus Buccal Misoprostol Alone for the Prevention of Postpartum Hemorrhage Following an Emergent Cesarean Delivery
Brief Title: Buccal Misoprostol and Intravenous Tranexamic Acid During Emergent Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: hany farouk (Other)
Responsible Party: Sponsor-Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu /185/18
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; tranexamic acid; postpartum hemorrhage; misoprostol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: A Double-Blind Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a double-blinded randomized placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Misoprostol with TA (Active Comparator): 400 μg of buccal misoprostol (two tablets) plus 1 gm tranexamic acid in 100 ml saline by iv rout
  Interventions: Drug: Misoprostol; Drug: TA
- Misoprostol with placebo to TA (Active Comparator): 400 μg of buccal misoprostol (two tablets) plus 110 ml saline by iv rout
  Interventions: Drug: Misoprostol; Drug: placebo to TA
- placebo to Misoprostol and TA (Placebo Comparator): placebo to misoprostol plus placebo to tranexamic acid
  Interventions: Drug: TA; Drug: placebo to misoprostol

INTERVENTIONS:
Drug: Misoprostol — 400 μg of buccal misoprostol
  Other Names: Active Comparator
  Arms: Misoprostol with TA; Misoprostol with placebo to TA
Drug: TA — 1 gm of tranexamic acid in 100 ml saline iv
  Other Names: active comparator
  Arms: Misoprostol with TA; placebo to Misoprostol and TA
Drug: placebo to misoprostol — placebo tablets to misoprostol buccal
  Other Names: Placebo comparator
  Arms: placebo to Misoprostol and TA
Drug: placebo to TA — 110 ml saline iv
  Other Names: placebo comparator
  Arms: Misoprostol with placebo to TA

SUMMARY:
Purpose to evaluate the effects of buccal misoprostol with or without intravenous tranexamic acid (TA) in comparison with placebo on reducing post-partum hemorrhage in pregnant women undergoing emergent cesarean section

DETAILED DESCRIPTION:
The American Congress of Obstetricians and Gynecologists (ACOG) defines postpartum hemorrhage (PPH) as the loss of more than 1,000 mL after cesarean delivery. In the majority of cases, uterine atony is responsible for the occurrence of excessive bleeding during or following childbirth. The Millennium Development Goal of reducing the maternal mortality ratio by 75 % by 2015 will remain beyond the investigator reach unless prioritize the prevention and treatment of PPH in low-resource countries. Consequently, the administration of uterotonic drugs during cesarean section (CS) has become essential to diminish the risk of PPH and improve maternal safety. Misoprostol is a prostaglandin E1 analog proven in several randomized controlled trials to be effective in preventing PPH because of its strong uterotonic effects. In addition, misoprostol is inexpensive, stable at room temperature, and easy to administer. Misoprostol has been broadly studied in the prevention and treatment of PPH after vaginal delivery; however, its use in conjunction with CS has not been investigated as much.T he buccal route is recognized as having the greatest benefit due to its rapid uptake, long-acting effect, and greatest bioavailability compared with other routes of misoprostol administration. Anti-fibrinolytic agents, such as tranexamic acid (TA), reduce the risk of death in bleeding trauma patients. On the other hand, it has been suggested that TA administration reduces blood loss and the incidence of PPH in females after vaginal or elective CS. The investigators designed this study to evaluate and compare these two new therapeutic options in controlling PPH following emergent CS.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years, singleton pregnancy, term gestation and decision made for a cesarean section in labor

Exclusion Criteria:

* multiple gestations
* placenta praevia and placental abruption
* undergoing cesarean section with general anesthesia
* women undergoing cesarean section at less than 37 weeks of gestation--with a severe medical disorder
* allergy to tranexamic acid or misoprostol
* refuse to consent
* elective cesarean section

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — age >18 years, singleton pregnancy, term gestation and decision made for a cesarean section in labor
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
estimation of intraoperative blood loss (ml) | during the operation
  measure Intraoperative blood loss in ml by gravimetric methods

SECONDARY OUTCOMES:
amount of postoperative blood loss | 6 hours post operative
  measure amount of blood loss post operative in ml by gravimetric methods
number of patient with postpartum hemorrhage | 24 hours post operative
  calculation of the number of the patients with blood loss >1000 ml

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided